CLINICAL TRIAL: NCT01708343
Title: Paraspinal Stimulation Combined With Trigger Point Needling and Needle Rotation in Treating Myofascial Pain: Randomized Sham-controlled Clinical Trial
Brief Title: Paraspinal Stimulation in Treating MPS
Acronym: DIMMST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, MD, PhD, Professor and coordinator of Pain & Neuromodulation Lab, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPS-DIMS
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Clinical Study - RCT
Keywords: Myofascial Pain Syndrome,; intramuscular stimulation,; acupuncture,; sleep quality,; pain threshold.
MeSH Terms: conditions — Myofascial Pain Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo-sham (Sham Comparator): Placebo-sham twice a week during four weeks
  Interventions: Procedure: DIMMST
- Lidocaine injection (Active Comparator): Lidocaine 0.2-0.5 mL of 1% injected each time into the trigger point. Twice a week during four weeks
  Interventions: Procedure: DIMMST
- DIMMST (Experimental): DIMMST include the combination of trigger point deep dry needling (TrP-DDN) is combined with paraspinal deep intramuscular stimulation (PDIMS) and needle rotation (NR).
  Twice a week during four weeks
  Interventions: Procedure: DIMMST

INTERVENTIONS:
Procedure: DIMMST
  Other Names: Eletroacupuncture; Myofascial pain

SUMMARY:
To test the hypothesis that the effect of either multiple deep intramuscular stimulation therapy [(DIMMST: trigger point deep dry needling (TrP-DDN) is combined with paraspinal deep intramuscular stimulation (PDIMS) and needle rotation (NR)] would be more effective than a placebo-sham for the treatment of MPS and that DIMMST would be more effective than LTrP-I for improving pain relief, sleep quality, and physical and mental state of the patient.

ELIGIBILITY:
Inclusion criteria

* Myofascial pain syndrome (MPS) (defined as regional pain, normal neurologic examination, presence of TrPs, taut bands, tender points, and pain characterized as "dull," "achy," or "deep" were relevant to MPS diagnosis. Additionally, palpable nodules, pain that is exacerbated by stress, decreased range of motion, and ropiness in the muscle).
* Disability in the last three months: (defined if they had one or more these limitation in active and routine activities by MPS : (i) interference with work, (ii) enjoyable activities, (iii) responsibilities at home, (iv) relationships, (v) personal goals, (vi) thinking clearly, and problem solving, concentrating, or remembering during the last three months).
* Women
* Age: 19 to 50 years

Exclusion criteria

Rheumatoid arthritis

Fibromyalgia

Previous surgery on the affected areas

Prior experience with acupuncture

Primary radiculopathy

Current use of psychotropic drugs (ilicits

) Habitual use of anti-inflammatory steroids.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Pain severity | A cumulative mean of each week during the treatmetn period (four weeks - the pain diary begin in the first of treatment to the last session)
  a) The intensity of pain was measured by a 10-cm VAS [30]. VAS scores ranged from no pain (zero) to the worst possible pain (10 cm).
Pain threshold | A cumulative mean of each week during the treatmetn period (four weeks - the pain diary begin in the first of treatment to the last session)
  Pain pressure threshold (PPT)

SECONDARY OUTCOMES:
Sleep quality - how did you feel when you woke up | A cumulative mean of each week during the treatmetn period (four weeks - the pain diary begin in the first of treatment to the last session)
  Sleep quality was recorded daily by the 10-cm visual analog sleep quality scale (VASQS) in the sleep diary using VASQS:
  In general, how did you feel when you woke up?
Sleep quality - compared to your habitual sleep | A cumulative mean of each week during the treatmetn period (four weeks - the pain diary begin in the first of treatment to the last session)
  Sleep quality was recorded daily by the 10-cm visual analog sleep quality scale (VASQS) in the sleep diary using VASQS:
  Assess the sleep quality of the previous night compared to your habitual sleep?
Sleep quality -last night | A cumulative mean of each week during the treatmetn period (four weeks - the pain diary begin in the first of treatment to the last session)
  Sleep quality was recorded daily by the 10-cm visual analog sleep quality scale (VASQS) in the sleep diary using VASQS:
  How well did you sleep last night?

OTHER OUTCOMES:
Physical and mental Health | Before to begin treatment and after end treatment
  Health-related quality of life, assessed at baseline and the end of treatment sessions, was measured with the SF-12 Summary Scales

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas E Porto Alegre, Porto Alegre, Rio Grande do Sul